CLINICAL TRIAL: NCT01027858
Title: Role of Exercise on Cognition and Function in Seniors With Vascular Cognitive Impairment: A Randomized Controlled Trial
Brief Title: PROMOTE: Promotion of the Mind Through Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Stroke Network (Other); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H09-00529
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Vascular Cognitive Impairment
Keywords: exercise; aerobic exercise training; vascular cognitive impairment; Mild Sub-cortical Ischaemic Vascular Cognitive Impairment (SIVCI)
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AT (aerobic-based exercise training)
  Interventions: Behavioral: Aerobic-based exercise training
- 2 (Active Comparator): CON (control; usual care)
  Interventions: Behavioral: CON (control; usual care)

INTERVENTIONS:
Behavioral: Aerobic-based exercise training — Six months of thrice-weekly walking program that will gradually progress in intensity. Each training session will be 60 minutes (10 minutes of warm-up, 40 minutes of training, and 10 minutes of cool-down).
  Arms: 1
Behavioral: CON (control; usual care) — Nutrition education and usual care as prescribed by neurologist
  Arms: 2

SUMMARY:
The investigators will conduct a proof-of-concept study to provide preliminary evidence of efficacy of aerobic-based exercise training for maintaining cognitive function, executive function, and everyday function in adults with mild vascular cognitive impairment.

DETAILED DESCRIPTION:
A total of 70 adults diagnosed with Ischaemic Vascular Cognitive Impairment (SIVCI) will be randomized to either a 6 month thrice weekly walking program or usual care. After 6 months of intervention, they will be followed for an additional 6 months. There will be three measurement sessions: baseline, 6 months (end of intervention period); and 12 months.

ELIGIBILITY:
Inclusion Criteria:

The study will specifically recruit individuals who fulfill the diagnostic criteria for SIVCI as outlined by Erkinjuntti and colleagues (1), which requires the presence of both cognitive syndrome (as defined in Section A below) and small vessel ischaemic disease (as defined in Section B below).

A. Cognitive Syndrome defined as:

1. Dysexecutive Syndrome: Some impairment in goal formulation, initiation, planning, organizing, sequencing, executing, set-shifting and maintenance, or abstracting.
2. Memory Deficit: Some impairment in recall, relative intact recognition, less severe forgetting, benefit from cues.
3. Progression: Deterioration of A1 and A2 from a previous higher level of functioning that are not per se interfering with complex occupational and social activities.

B. Small Vessel Ischaemic Disease defined as:

1. Evidence of relevant cerebrovascular disease by brain imaging (in the last 12 months) defined as the presence of both:

   i. Periventricular and deep white matter lesions: Patchy areas of low attenuation (intermediate density between that of normal white matter and that of intraventricular cerebro-spinal fluid) or diffuse symmetrical areas of low attenuation with ill defined margins extending to the centrum semiovale plus at least one lacunar infarct (correlating to the white matter grading scale greater than 3 from the Cardiovascular Health Study) (2,3); and ii. Absence of cortical and/or cortico-sub-cortical non-lacunar territorial infarcts and watershed infarcts, haemorrhages indicating large vessel disease, signs of normal pressure hydrocephalus, or other specific causes of white matter lesions (e.g., multiple sclerosis, leukodystrophies, sarcoidosis, brain irradiation, etc).
2. Presence or a history of neurological signs as evidence for cerebrovascular disease such as hemiparesis, lower facial weakness, Babinski sign, sensory deficit, dysarthria, gait disorder, extrapyramidal signs consistent with sub-cortical brain lesion(s).

In addition, individuals must meet the following inclusion criteria:

1. Montreal Cognitive Assessment (MoCA) (4) score less than 26 at screening;
2. MMSE (5) score of > 20 at screening;
3. Community-dwelling;
4. Lives in Metro Vancouver;
5. Have a caregiver, family member, or friend who interacts with him/her on a weekly basis;
6. Able to comply with scheduled visits, treatment plan, and other trial procedures;
7. Must be able to read, write, and speak English in which psychometric tests are provided with acceptable visual and auditory acuity;
8. Stable on a fixed dose of cognitive medications (e.g., donepezil, galantamine, rivastigmine, memantine, etc.) that is not expected to change during the 12-month study period, or, if they are not on any of these medications, they are not expected to start them during the 12-month study period;
9. Provide a personally signed and dated informed consent document indicating that the individual (or a legally acceptable representative) has been informed of all pertinent aspects of the trial. In addition, an assent form will be provided at baseline and again at regular intervals;
10. Able to walk independently; and
11. Must be in sufficient health to participate in study's aerobic-based exercise training program. This will be based on medical history, vital signs, physical examination by study physicians, and written recommendation by family physician indicating individual's appropriateness to participate in an aerobic-based exercise training program.

Exclusion Criteria:

1. Absence of relevant small vessel ischaemic lesions on an existing brain computed tomography (CT) or MRI;
2. Diagnosed with another type of dementia (e.g., AD) or other neurological conditions (e.g., multiple sclerosis, Parkinson's disease, etc.) that affects cognition and mobility;
3. At high risk for cardiac complications during exercise and/or unable to self-regulate activity or to understand recommended activity level (i.e., Class C of the American Heart Risk Stratification Criteria);
4. Have clinically significant peripheral neuropathy or severe musculoskeletal or joint disease that impairs mobility;
5. Taking medications that may negatively affect cognitive function, such as anticholinergics, including agents with pronounced anticholinergic properties (e.g., amitriptyline), major tranquilizers (typical and atypical antipsychotics), and anticonvulsants (e.g., gabapentin, valproic acid, etc.); or
6. Individual who plans to participate or is enrolled in a clinical drug trial concurrent to this study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
This is a proof-of-concept study. The primary endpoints are: ADAS-Cog | baseline, 6 months, and 12 months
EXIT-25 | baseline, 6 months, and 12 months
ADCS-ADL | baseline, 6 months, and 12 months

SECONDARY OUTCOMES:
Secondary outcomes of interest include: performance of specific executive processes | baseline, 6 months, and 12 months
Physical function | baseline, 6 months, and 12 months
Inflammatory biomarkers | baseline, 6 months, and 12 months
Serum glucose and lipids. These will be assessed at 6 and 12 months. | baseline, 6 months, and 12 months

OTHER OUTCOMES:
Brain Structure | Baseline and 6 months
  Volume and white matter lesions.
Brain Function | Baseline and 6 months
  fMRI and resting state

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, Ph.D, PT, Principal Investigator — University of British Columbia; Janice Eng, Ph.D, Study Director — University of British Columbia; Lara Boyd, Ph.D, Study Director — University of British Columbia; Robin Hsiung, Ph.D, Study Director — University of British Columbia; Claudia Jacova, Ph.D, Study Director — University of British Columbia; Howard Feldman, MD, Study Director — University of British Columbia; Penny Brasher, Ph.D, Study Director — University of British Columbia; Philip Lee, Ph.D, Study Director — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Liu-Ambrose T, Best JR, Davis JC, Eng JJ, Lee PE, Jacova C, Boyd LA, Brasher PM, Munkacsy M, Cheung W, Hsiung GR. Aerobic exercise and vascular cognitive impairment: A randomized controlled trial. Neurology. 2016 Nov 15;87(20):2082-2090. doi: 10.1212/WNL.0000000000003332. Epub 2016 Oct 19. PMID 27760869
- [Background] Liu-Ambrose T, Eng JJ, Boyd LA, Jacova C, Davis JC, Bryan S, Lee P, Brasher P, Hsiung GY. Promotion of the mind through exercise (PROMoTE): a proof-of-concept randomized controlled trial of aerobic exercise training in older adults with vascular cognitive impairment. BMC Neurol. 2010 Feb 17;10:14. doi: 10.1186/1471-2377-10-14. PMID 20158920
- [Background] Hsu CL, Best JR, Davis JC, Nagamatsu LS, Wang S, Boyd LA, Hsiung GR, Voss MW, Eng JJ, Liu-Ambrose T. Aerobic exercise promotes executive functions and impacts functional neural activity among older adults with vascular cognitive impairment. Br J Sports Med. 2018 Feb;52(3):184-191. doi: 10.1136/bjsports-2016-096846. Epub 2017 Apr 21. PMID 28432077
- [Background] Barha CK, Hsiung GR, Best JR, Davis JC, Eng JJ, Jacova C, Lee PE, Munkacsy M, Cheung W, Liu-Ambrose T. Sex Difference in Aerobic Exercise Efficacy to Improve Cognition in Older Adults with Vascular Cognitive Impairment: Secondary Analysis of a Randomized Controlled Trial. J Alzheimers Dis. 2017;60(4):1397-1410. doi: 10.3233/JAD-170221. PMID 29036816
- [Background] Dao E, Barha CK, Best JR, Hsiung GY, Tam R, Liu-Ambrose T. The Effect of Aerobic Exercise on White Matter Hyperintensity Progression May Vary by Sex. Can J Aging. 2019 Jun;38(2):236-244. doi: 10.1017/S0714980818000582. Epub 2019 Mar 14. PMID 30867079
- [Background] A history of the Arkansas State Dental Hygienists Association. Ark Dent J. 1987 Apr;58(1):43. No abstract available. PMID 3107531
- [Background] Barha CK, Dao E, Marcotte L, Hsiung GR, Tam R, Liu-Ambrose T. Cardiovascular risk moderates the effect of aerobic exercise on executive functions in older adults with subcortical ischemic vascular cognitive impairment. Sci Rep. 2021 Oct 7;11(1):19974. doi: 10.1038/s41598-021-99249-1. PMID 34620933
- [Derived] Barha CK, Starkey SY, Hsiung GYR, Tam R, Liu-Ambrose T. Aerobic exercise improves executive functions in females, but not males, without the BDNF Val66Met polymorphism. Biol Sex Differ. 2023 Apr 3;14(1):16. doi: 10.1186/s13293-023-00499-7. PMID 37013586
- [Derived] Barha CK, Hsiung GYR, Liu-Ambrose T. The Role of S100B in Aerobic Training Efficacy in Older Adults with Mild Vascular Cognitive Impairment: Secondary Analysis of a Randomized Controlled Trial. Neuroscience. 2019 Jul 1;410:176-182. doi: 10.1016/j.neuroscience.2019.04.052. Epub 2019 May 7. PMID 31075314
- [Derived] Dao E, Best JR, Hsiung GR, Sossi V, Jacova C, Tam R, Liu-Ambrose T. Associations between cerebral amyloid and changes in cognitive function and falls risk in subcortical ischemic vascular cognitive impairment. BMC Geriatr. 2017 Jun 28;17(1):133. doi: 10.1186/s12877-017-0522-4. PMID 28659161
- [Derived] Davis JC, Hsiung GR, Bryan S, Best JR, Eng JJ, Munkacsy M, Cheung W, Chiu B, Jacova C, Lee P, Liu-Ambrose T. Economic evaluation of aerobic exercise training in older adults with vascular cognitive impairment: PROMoTE trial. BMJ Open. 2017 Mar 29;7(3):e014387. doi: 10.1136/bmjopen-2016-014387. PMID 28360247
- [Derived] Davis JC, Hsiung GY, Bryan S, Jacova C, Jacova P, Munkacsy M, Cheung W, Lee P, Liu-Ambrose T. Agreement between Patient and Proxy Assessments of Quality of Life among Older Adults with Vascular Cognitive Impairment Using the EQ-5D-3L and ICECAP-O. PLoS One. 2016 Apr 21;11(4):e0153878. doi: 10.1371/journal.pone.0153878. eCollection 2016. PMID 27101402
- [Derived] Dao E, Hsiung GY, Sossi V, Jacova C, Tam R, Dinelle K, Best JR, Liu-Ambrose T. Exploring the effects of coexisting amyloid in subcortical vascular cognitive impairment. BMC Neurol. 2015 Oct 12;15:197. doi: 10.1186/s12883-015-0459-1. PMID 26459220